CLINICAL TRIAL: NCT03039140
Title: A Cardiac Rehabilitation Program for Breast Cancer Survivors: A Feasibility Study
Brief Title: Cardiac Rehabilitation Program in Improving Cardiorespiratory Fitness in Stage 0-III Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-14060; NCI-2015-00810 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-03-07; First posted 2017-02-01 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Cancer Survivor; Stage 0 Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (CR program) (Experimental): Patients participate in a CR program consisting of 1-hour CR intervention sessions, based on a personalized exercise prescription, 3 times per week for 14 weeks (a total of 36 sessions). Components of the exercise prescription includes intensity, mode, duration, and frequency. Intensity of exercise is guided by the results of a graded exercise stress test, RPE, heart rate, and symptoms, such as chest pain/angina or shortness of breath. If exercise is well-tolerated during CR sessions, patients are encouraged to supplement their exercise program at home, increasing their exercise frequency to up to 5 times per week. Patients may attend weekly educational sessions offered by the Phase 2 CR program which covers topics such as stress management, smoking cessation, nutrition, and weight loss.
  Interventions: Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Attend weekly educational sessions
  Other Names: Education for Intervention; Intervention, Educational
Behavioral: Exercise Intervention — Participate in CR program
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies a cardiac rehabilitation program in improving cardiorespiratory fitness in stage 0-III breast cancer survivors. Cardiovascular disease is the leading cause of death of women in both the general population and the breast cancer survivor population. There are many risk factors common to both heart disease and breast cancer development, including physical inactivity. A cardiac rehabilitation program may help improve cardiorespiratory fitness, reduce cardiovascular disease risk factors, and improve quality of life among breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility of conducting a 14-week cardiac rehabilitation (CR) program in women with breast cancer after completion of acute therapy.

II. Preliminarily evaluate the efficacy of CR in improving cardiorespiratory fitness (peak oxygen uptake, maximum volume of oxygen [VO2 max]) at baseline and 14 weeks.

III. Explore changes in cardiovascular disease (CVD) risk factors (blood pressure, cholesterol, fasting glucose, and body mass index) between baseline and 14-week follow-up. Blood pressure and body mass index will also be checked at 8 weeks.

IV. Quantify the difference in quality of life (QoL) between baseline, 8 week, and 14 week follow up, adjusting for baseline QoL values.

OUTLINE:

Patients participate in a CR program consisting of 1-hour CR intervention sessions, based on a personalized exercise prescription, 3 times per week for 14 weeks (a total of 36 sessions). Components of the exercise prescription includes intensity, mode, duration, and frequency. Intensity of exercise is guided by the results of a graded exercise stress test, rating of perceived exertion (RPE), heart rate, and symptoms, such as chest pain/angina or shortness of breath. If exercise is well-tolerated during CR sessions, patients are encouraged to supplement their exercise program at home, increasing their exercise frequency to up to 5 times per week. Patients may attend weekly educational sessions offered by the Phase 2 CR program which covers topics such as stress management, smoking cessation, nutrition, and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer stages 0-III within 6 months after completion of all planned surgery, radiation and or chemotherapy treatments
* Concurrent endocrine therapy permissible
* Ability to understand and the willingness to sign a written informed consent
* Willingness to participate in CR program

Exclusion Criteria:

* Existing CVD
* Existing diabetes
* Contraindications to exercise
* Metastatic breast cancer
* Other concurrent malignancies except skin cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnant or nursing women
* Unable to give informed consent
* Any contraindication to cardiac stress testing
* Travel distance greater than 50 miles

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a 14-week CR program | 14 weeks
  During the course of the 14-week intervention period, the CR medical director will monitor CR staff adherence to the study protocol. Every 2 weeks, they will review intervention participants' baseline graded exercise test results and subsequent exercise prescriptions to ensure the intervention is targeted at the appropriate level of each participant's VO2 max. Will administer a satisfaction questionnaire to intervention participants. Results from these surveys will be evaluated during the course of the study by the principal investigator and used to improve the study process as appropriate.

SECONDARY OUTCOMES:
Efficacy of CR in improving cardiorespiratory fitness | At 14 weeks
  Analysis of follow-up VO2 max, in units of mL/kg/min, will be done using an analysis of covariance (ANCOVA) approach. If VO2 max values are missing at 14 weeks, will use the Duke Activity Status Index questionnaire responses to approximate VO2 max values.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Lustberg, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu